CLINICAL TRIAL: NCT02997150
Title: Treatment of Steroid Dependent Idiopathic Nephrotic Syndrome in Children With Low Doses of Interleukin 2: a Pilot Study
Acronym: NIL-2 pilote
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no treatment available
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I15041 (NIL-2 pilote)
Record Dates: First submitted 2016-12-15; First posted 2016-12-19 (Estimated); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Nephrotic Syndrome Steroid-Dependent; Interleukin 2
Keywords: Idiopathic nephrotic syndrome-child-steroid dependant-IL2; Safety; Efficacy
MeSH Terms: conditions — Nephrotic Syndrome | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IL-2 low dose (Experimental)
  Interventions: Drug: IL-2 Low dose

INTERVENTIONS:
Drug: IL-2 Low dose — Patients receive low doses of Interleukin 2: 0.5 million UI/m²/ injection subcutaneously.
  The treatment is initiated with an induction phase of one injection per day for 5 consecutive days, followed by a maintenance phase in which patients will receive one injection every 14 days for 6 months.
  At the same time, corticoid treatment will be tapered until its complete withdrawal no later than 3 months from the first injection

SUMMARY:
NIL-2 is a clinical trial designed to evaluate the efficacy and safety of low doses of Interleukin2 in the treatment of recently diagnosed, steroid dependent idiopathic nephrotic syndrome in children. Recent data suggest that Interleukin 2 could be an effective therapy via an increased production of regulatory T cells.

DETAILED DESCRIPTION:
The study will include 10 children (age: 3-15 years old). Patients will receive low doses of Interleukin 2 (0.5 million UI/m²/ injection, subcutaneously).

The treatment will be initiated with an induction phase of one injection per day for 5 consecutive days, followed by a maintenance phase in which patients will receive one injection every 14 days for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 15 years of age (included) with a steroid responsive idiopathic nephrotic syndrome
* Idiopathic nephrotic syndrome progressing for less than 1 year
* Steroid dependent idiopathic nephrotic syndrome (at least 1 relapse when steroids are tapered off or within 3 months after their withdrawal, and reliance on steroids > 15 mg/m² every other day)
* Steroid dose at inclusion between 15 and 60 mg/m²every other day
* Patient with a stable dose of steroids within the 8 days before and after the first injection of IL2
* Patient in remission for more than 15 days
* Patient affiliated to a French health insurance
* Signed consent of parental authority

Exclusion Criteria:

* Hypersensitivity to IL2 or to one of its excipients
* Significant history or presence of cardiopathy
* Signs of evolving infection requiring an antibiotic treatment
* Respiratory distress, respiratory infection or chronic respiratory failure
* Serious dysfunction of one of the vital organs
* Leukocytes < 4000/mm3 ; platelets < 100 000/mm3; hematocrit <30%
* Anomaly of serum bilirubin and creatinin levels
* History of organ allograft
* Other pre-existing autoimmune disease
* Male and female pubescent teenagers under the age of 15
* Male and female teenagers whose puberty has begun for more than one year
* Asthmatic patient
* Pregnant or breastfeeding female patient
* Participation in another therapeutic trial concurrently or 30 days prior to inclusion

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-02 (Estimated); Primary Completion 2018-08 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Number of success: absence of relapse of idiopathic nephrotic syndrome | Day 184
  Absence of relapse of idiopathic nephrotic syndrome

SECONDARY OUTCOMES:
Safety of Interleukin-2 | Day 214
  Study of adverse events
Increase of regulatory T cells after 5 injections of Interleukin-2 | Day 8
  increase of regulatory T cells (CD4+, CD25+, Foxp3 cells) from baseline to fifth injection, expressed as a percentage
Increase of regulatory T cells after 18 injections of Interleukin-2 | Day 184
  increase of regulatory T cells (CD4+, CD25+, Foxp3 cells) from baseline to eighteenth injection, expressed as a percentage

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Guigonis, MD, Principal Investigator — University Hospital, Limoges